CLINICAL TRIAL: NCT04473742
Title: Effects of Silica and Asbestos Fibres on the Efferocytosis Capacities of Macrophages
Acronym: MacFibOsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC20_8878_MacFibOsis
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: History of Exposure to Silica or Asbestosis; Positive Testing for ANA as a Marker of Systemic Autoimmune Diseases
Keywords: efferocytosis; macrophages; silica; asbestosis; HMGB1; osteopontin
MeSH Terms: conditions — Asbestosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients exposed to silica (Experimental)
  Interventions: Biological: Blood collection; Biological: Blood sample
- Patients exposed to asbestos fibres (Active Comparator)
  Interventions: Biological: Blood collection; Biological: Blood sample

INTERVENTIONS:
Biological: Blood collection — 4 EDTA tubes for 24 mL blood collection
Biological: Blood sample — 2 drying tubes for 12 mL blood collection
  Arms: Patients exposed to asbestos fibres
Biological: Blood sample — 1 drying tube for 6 mL blood collection
  Arms: Patients exposed to silica

SUMMARY:
Evaluation of the efferocytosis capacities of blood Monocyte Derived Macrophages (MDM) from patients with a history of asbestosis or silica exposure and comparison of these capacities with those of MDM from healthy donors.

DETAILED DESCRIPTION:
Patients with a proven history or current exposure will have 4 EDTA tubes drawn, approximately 24mL of fresh whole blood for efferocytosis assessment and :

* 2 x 6mL serum tubes for the assessment of Antinuclear Antibody (ANA) positivity, serum high-mobility group box 1 (HMGB1) and osteopontin for patients exposed to asbestos
* 1 x 6mL serum tube for serum HMGB1 and osteopontin for patients exposed to silica

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 Yo
* Addressed to the department of occupational disease
* With a history of asbestosis or silica exposure evaluated by a dedicated questionnaire and a throughout examination of the history of occupations, according to standard procedures for the follow-up of at risk workers.
* Persons who received an oral and written information on the protocol and signed the informed consent form

Exclusion Criteria:

* Pregnant or breastfeeding women
* Subject legally protected (under judicial protection, guardianship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Efferocytosis Index (EI) calculation (%) defined as the number of efferocyte MDM / total number of MDM | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
EI calculation in patients positive for ANA vs patients negative for ANA | Through study completion, an average of 2 years
Serum concentration of HMGB1 and Osteopontin (SPP1) by ELISA | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No